CLINICAL TRIAL: NCT01973595
Title: Almonds: Digestive Health and Immune Function of Adults and Children: a Randomized Crossover Study
Brief Title: Almonds: Digestive Health and Immune Function of Adults and Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Almond Board of California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 201300475
Record Dates: First submitted 2013-10-15; First posted 2013-10-31 (Estimated); Results first posted 2016-04-25 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: almonds; inflammation; immunity; gut microbiota; stress; diet quality
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Almonds then no almonds (Experimental): Adults will consume 1.5 ounces of almonds or almond paste per day and children will consume 0.5 ounces of almonds or almond paste per day for 3 weeks.
  Interventions: Dietary Supplement: Almonds, Then no almonds
- No almonds then almonds (Other): No almonds will be consumed by participants for 3 weeks.
  Interventions: Other: No Almonds, Then almonds

INTERVENTIONS:
Dietary Supplement: Almonds, Then no almonds — Whole, raw almonds with skin, or whole, raw almonds with skin that have been ground into a paste.
  Arms: Almonds then no almonds
Other: No Almonds, Then almonds — No almonds will be consumed by participants for 3 weeks.
  Arms: No almonds then almonds

SUMMARY:
The purpose of this study is to determine whether incorporating almonds into the diets of families with young children will induce beneficial changes in gastrointestinal function, the fecal microbiota profile, and immune and inflammatory processes of the adults and children resulting in improved quality of life. The investigators anticipate finding an increase in beneficial bacteria, improved intestinal function, and decreased inflammation during the almond intervention.

DETAILED DESCRIPTION:
This is a randomized, crossover study. After obtaining informed consent, healthy adults aged 18-40 years with children aged 3-6 years will be randomized to either consume almonds and almond paste during the first arm of the study or during the second arm of the study. During the intervention period, adult participants will consume 1.5 ounces of almonds per day, and children will consume 0.5 ounces of almonds per day for 3 weeks. After a 4-week washout period, participants will be crossed to the other treatment (no almond consumption or almond consumption).

Participants will complete daily questionnaires throughout the intervention period, and one week before and after each intervention period. Blood samples will be collected from adults at the baseline and final time points of each intervention. Stool samples will be collected during the pre-baseline and final weeks of each intervention. Dietary intake will be assessed weekly during each intervention period. Gastrointestinal symptoms questionnaires will be completed weekly during each intervention.

ELIGIBILITY:
Inclusion Criteria:

To participate in the study, adult participants must:

* Be 18 to 40 years old.
* Have a 3 to 6 year old child that you are willing to enroll in the study.
* Live with your child for on average at least 6 days of the week.
* Be willing and able to complete the Informed Consent Form in English.
* Not be currently pregnant or planning to become pregnant in the next 5 months.
* Be willing to consume 1.5 ounces of almonds (~43 nuts) each day for three weeks.
* Be willing to feed your child 0.5 ounces of almond paste (~2 tablespoons) per day for three weeks.
* Be willing monitor your child's daily intake over the course of the study.
* Be willing to provide 4 blood samples, 4 stool samples, and 4 saliva samples over the course of the study.
* Be willing to assist your child in providing 4 stool samples and 4 saliva samples over the course of the study.
* Be willing and able to complete daily and weekly questionnaires for you and your child regarding general wellness, bowel function, gastrointestinal symptoms, stress and anxiety, and dietary intake.
* Must be available for 14 consecutive weeks to participate in the study.

Exclusion Criteria:

To participate in the study, adult and child participants:

* Must not have any known nut or tree nut allergies.
* Must discontinue any immune-enhancing dietary supplements (e.g., prebiotics and fiber supplements, probiotics, fish oil, vitamin E >400% of the Recommended Dietary Allowance (RDA) or >60 mg/day, and yogurts with live, active cultures).
* Must not be currently taking any medications for constipation or diarrhea on a regular basis.
* Must not be currently taking any large doses of anti-inflammatory drugs (i.e., aspirin in doses >600 mg/d) on a regular basis.
* Must not have received antibiotic therapy or a colonoscopy in the past two months.
* Must not be currently being treated for or have any of the following physician-diagnosed diseases or conditions: HIV/AIDS; immune modulating diseases (autoimmune disease, hepatitis, cancer); kidney disease; pancreatitis; pulmonary disease; hepatic or biliary disease; or gastrointestinal diseases/conditions such as diverticulitis, ulcerative colitis, Crohn's disease, Celiac disease, short bowel disease, ileostomy, or colostomy, but not including gastroesophageal reflux disease; or have a central venous catheter.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2013-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bobbi Langkamp-Henken, PhD, RD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] Burns AM, Zitt MA, Rowe CC, Langkamp-Henken B, Mai V, Nieves C Jr, Ukhanova M, Christman MC, Dahl WJ. Diet quality improves for parents and children when almonds are incorporated into their daily diet: a randomized, crossover study. Nutr Res. 2016 Jan;36(1):80-9. doi: 10.1016/j.nutres.2015.11.004. Epub 2015 Nov 10. PMID 26773784

RESULTS

PARTICIPANT FLOW:
Groups:
- Almonds, Then no Almonds (Parents): Parents were asked to consume 1.5 ounces of almonds or almond paste per day for 3 weeks. After a washout period of 4 weeks, they then received control diet.
  Almonds: Whole, raw almonds with skin, or whole, raw almonds with skin that have been ground into a paste.
- No Almonds, Then Almonds (Parents): Parents were asked not to consume almonds for 3 weeks. After a washout period of 4 weeks, they then received the almond intervention diet.
- Almonds, Then no Almonds (Children): Children were asked to consume 0.5 ounces of almonds or almond paste per day for 3 weeks. After a washout period of 4 weeks, they then received control diet.
  Almonds: Whole, raw almonds with skin, or whole, raw almonds with skin that have been ground into a paste.
- No Almonds Then Almonds (Children): Children were asked not to consume almonds for 3 weeks. After a washout period of 4 weeks, they then received the almond intervention diet.
Period: Intervention Phase 1
Arm/Group | Almonds, Then no Almonds (Parents) | No Almonds, Then Almonds (Parents) | Almonds, Then no Almonds (Children) | No Almonds Then Almonds (Children)
Started | 15 | 14 | 15 | 14
Completed | 15 | 14 | 15 | 14
Not Completed | 0 | 0 | 0 | 0
Period: Washout
Arm/Group | Almonds, Then no Almonds (Parents) | No Almonds, Then Almonds (Parents) | Almonds, Then no Almonds (Children) | No Almonds Then Almonds (Children)
Started | 15 | 14 | 15 | 14
Completed | 14 | 14 | 14 | 14
Not Completed | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Period: Intervention Phase 2
Arm/Group | Almonds, Then no Almonds (Parents) | No Almonds, Then Almonds (Parents) | Almonds, Then no Almonds (Children) | No Almonds Then Almonds (Children)
Started | 14 | 14 | 14 | 14
Completed | 14 | 14 | 14 | 14
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data from parents and children were analyzed separately. All parents and children received both treatments arms.
Groups:
- No Almonds, Then Almonds (Children): Children were asked not to consume almonds for 3 weeks. After a washout period of 4 weeks, they then received the almond intervention diet.
- Total: Total of all reporting groups
Arm/Group | Almonds, Then no Almonds (Parents) | No Almonds, Then Almonds (Parents) | Almonds, Then no Almonds (Children) | No Almonds, Then Almonds (Children) | Total
Number analyzed (Participants) | 15 | 14 | 15 | 14 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 15 | 14 | 29
  Between 18 and 65 years | 15 | 14 | 0 | 0 | 29
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 9 | 5 | 38
  Male | 2 | 3 | 6 | 9 | 20
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 15 | 14 | 58

OUTCOME MEASURES:

1. Primary Outcome: Gut Microbiota Community Composition
Description: The mean of the change between baseline and final time points in stool lactic acid bacteria counts [log(CFU)] was compared for each study arm.
Time Frame: Baseline #1 (Week 1) to Final #1 (Week 4) of each intervention
Population: Stool samples were analyzed only if all 4 were available from each participant. Therefore, only data from 21 parents and 20 children were analyzed.
Measure: Mean (Standard Error); unit: log (CFU)
Groups:
- Almonds Consumption: Participants were asked to consume 1.5 ounces of almonds or almond paste per day for 3 weeks.
  Each group received the almond intervention and the no almond consumption control.
  Almonds: Whole, raw almonds with skin, or whole, raw almonds with skin that have been ground into a paste.
- No Almonds Consumption Control: Participants were asked not to consume almonds for 3 weeks.
  Each group received the almond intervention and the no almond consumption control.
Arm/Group | Almonds Consumption | No Almonds Consumption Control
Number analyzed (Participants) | 41 | 41
log (CFU)
  Parents | -.0116 (0.162) | -0.407 (0.137)
  Children | -0.161 (0.292) | -.0498 (0.231)

2. Secondary Outcome: Inflammatory Status
Description: Levels of inflammatory markers in the blood (IL-6) were compared between baseline and final time points once the participants were on the Almonds intervention.. The data were collected at Baseline and Week four.
Time Frame: Change between Baseline to Week 4
Population: Parents (Almonds baseline, n=29, final n=29, No almonds baseline n=28, final n= 28; one parent withdrew prior to no almond consumption control intervention) were analyzed for almonds and no almond consumption, no children were included in this analysis.
Measure: Mean (Standard Error); unit: ng/ml
Groups:
- Almonds Consumption (Parents): Parents were asked to consume 1.5 ounces of almonds or almond paste per day for 3 weeks.
  Each group received the almond intervention and the no almond consumption control.
  Almonds: Whole, raw almonds with skin, or whole, raw almonds with skin that have been ground into a paste.
- No Almonds Consumption Control (Parents): Parents were asked not to consume almonds for 3 weeks.
  Each group received the almond intervention and the no almond consumption control.
Arm/Group | Almonds Consumption (Parents) | No Almonds Consumption Control (Parents)
Number analyzed (Participants) | 29 | 28
ng/ml
  Baseline | 13 (0.9) | 14 (0.9)
  Final | 14 (0.9) | 14 (0.9)

3. Secondary Outcome: Gastrointestinal Function
Description: Changes in average number of stools per week were measured using a Daily Questionnaire. Results were compared between treatment periods for each subject/group.
Time Frame: Pre-baseline (Week 0) and Week 3 of each intervention
Population: 29 parents and 29 children consumed almonds n=58; one parent-child pair withdrew prior to no almond consumption control intervention n=56; parents and children were analyzed for almonds and no almond consumption.
Measure: Mean (Standard Error); unit: average stools per week
Groups:
- No Almond Consumption Control: Participants were asked not to consume almonds for 3 weeks. After a washout period of 4 weeks, they then received the almond intervention diet.
  Each group received the almond intervention and the no almond consumption control.
Arm/Group | Almonds Consumption | No Almond Consumption Control
Number analyzed (Participants) | 58 | 56
average stools per week
  Parents Pre-baseline | 9.4 (0.8) | 8.6 (0.8)
  Parents Week 3 | 9.6 (0.8) | 10.3 (0.8)
  Children Pre-baseline | 6.7 (6.7) | 6.1 (0.5)
  Children Week 3 | 7.4 (0.5) | 6.9 (0.5)

4. Secondary Outcome: Diet Quality
Description: Three dietary recalls occurred per study arm, and each recall was scored for quality. The quality scores were averaged per arm and then compared between study arms for each subject/group using the Healthy Eating Index-2010.The Healthy Eating Index assesses diet quality based on 12 components, when summed has maximum points of 100 (HEI scale 0-100).
  High component scores indicate intakes close to the recommended ranges or amounts; low component scores indicate less compliance with the recommended ranges or amounts.
  National averages total score: children: 54.9 [4-8 years] and adults: 57.4 [31-50 years])
Time Frame: Three week almond intervention vs. three week no almond intervention
Population: 29 Parents and 29 children were analyzed separately for almonds and no almond consumption; one parent-child pair withdrew prior to no almond consumption control.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Almonds Consumption (Children): Children were asked to consume 0.5 ounces of almonds or almond paste per day for 3 weeks.
  Each group received the almond intervention and the no almond consumption control.
  Almonds: Whole, raw almonds with skin, or whole, raw almonds with skin that have been ground into a paste.
- No Almonds Consumption Control (Children): Children were asked not to consume almonds for 3 weeks.
  Each group received the almond intervention and the no almond consumption control.
Arm/Group | Almonds Consumption (Parents) | No Almonds Consumption Control (Parents) | Almonds Consumption (Children) | No Almonds Consumption Control (Children)
Number analyzed (Participants) | 29 | 28 | 29 | 28
units on a scale | 61.4 (1.4) | 53.7 (1.8) | 61.4 (2.2) | 53.7 (2.6)

ADVERSE EVENTS:
Time Frame: 14 weeks; pre-baseline (week 0) to final follow up week (week 14)
Arm/Group | Almonds Consumption | No Almonds Consumption Control
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/58
Other Adverse Events (participants affected / at risk) | 0/58 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No